CLINICAL TRIAL: NCT03727009
Title: Blood Sample Collection to Evaluate Biomarkers in Subjects With Untreated Hematologic Malignancies
Status: Terminated | Type: Observational
Why Stopped: COVID-19
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-02
Record Dates: First submitted 2018-10-23; First posted 2018-11-01 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Hematologic Malignancy
Keywords: blood draw; sample collections
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hematologic Malignancy: Subjects with clinically confirmed hematologic malignancy and who are treatment naive will provide a blood sample at the time of enrollment. No additional blood draws will occur.
  Interventions: Other: Blood Sample Collection

INTERVENTIONS:
Other: Blood Sample Collection — Subjects participating in the study will have blood drawn at enrollment.

SUMMARY:
The primary objective of this study is to obtain de-identified, clinically characterized, whole blood specimens to evaluate biomarkers associated with cancer for diagnostic assay development.

DETAILED DESCRIPTION:
Subjects will have been recently diagnosed with an untreated hematologic malignancy. Subjects will have a blood sample collected at enrollment and provide medical history prior to initiation of treatment. There will be no further follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female ≥ 18 years of age.
* Subject has an untreated hematologic malignancy.
* Subject understands the study procedures and is able to provide informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

* Any previous cancer diagnosis within the past 5 years (with the exceptions of basal cell or squamous cell skin cancers).
* Chemotherapy and/or radiation therapy within 5 years prior to enrollment/sample collection.
* Any treatment for the primary malignancy. Subject may not have started neo-adjuvant chemotherapy, neo-adjuvant radiation therapy, immunotherapy or other treatment prior to blood sample collection.
* Less than 3 days between fine needle aspiration (FNA) of target pathology and blood collection.
* Less than 7 days between biopsy (other than FNA) of target pathology and blood collection.
* IV contrast (e.g. CT and MRI) within 1 day [or 24 hours] of blood collection.
* Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 500 subjects will be enrolled. Subjects will be men and women, 18 years of age and older, who have an untreated hematologic malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Blood-based biomarkers associated with genetic and epigenetic alterations. | Point in time blood collection (1 day) at enrollment
  Biomarkers under evaluation include differential methylation of nucleic acids and altered expression of proteins in blood from subjects with a hematologic malignancy at the pre-intervention stage.

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Mercy Fort Smith, Fort Smith, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - Marin Cancer Care, Greenbrae, California
  - Alliance Research Centers, Laguna Hills, California
  - North County Oncology, Oceanside, California
  - Middlesex Hospital, Middletown, Connecticut
  - The Stamford Hospital, Stamford, Connecticut
  - Mid-Florida Hematology and Oncology Center, Orange City, Florida
  - PMG Research, INC, Downers Grove, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Orchard Healthcare Research, Inc., Skokie, Illinois
  - Carle Cancer Center NCI, Urbana, Illinois
  - Indiana Blood and Marrow Transportation, Indianapolis, Indiana
  - St. Elizabeth Medical Center, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - RCCA MD Inc., Bethesda, Maryland
  - Cancer Research Consortium of West Michigan, Grand Rapids, Michigan
  - HealthPartner Institute, Bloomington, Minnesota
  - Mercy Joplin, Joplin, Missouri
  - Mercy Springfield, Springfield, Missouri
  - Mercy St. Louis, St Louis, Missouri
  - East Carolina University Brody School of Medicine, Greenville, North Carolina
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - Mercy Oklahoma City, Oklahoma City, Oklahoma
  - Bon Secours St Francis Cancer Center, Greenville, South Carolina
  - Spartanburg Regional Healthcare District, Spartanburg, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Community Cancer Trials of Utah, Ogden, Utah
  - Wenatchee Valley Hospital, Wenatchee, Washington
  - CAMC Clinical Trials Center, Charleston, West Virginia
  - Dean Clinic - Fort Atkinson Specialty Services, Fort Atkinson, Wisconsin
  - ProHealth Care, Oconomowoc, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study will be shared after deidentification. This may include text, tables, figures, and appendices. The study protocol and informed consent form (when applicable) will also be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available from 2 years and ending 4 years after publication. Data will be shared with researchers who provide a methodologically sound proposal to achieve the aims outlined in the approved proposal.
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary IRB/EC approvals or waivers as applicable to conduct research. Data will be available between 2 and 4 years after publication through the Sponsor.